CLINICAL TRIAL: NCT02234973
Title: Transformation of Indigenous Primary Healthcare Delivery (FORGE AHEAD): Community-driven Innovations and Strategic Scale-up Toolkits
Brief Title: Transformation of Indigenous Primary Healthcare Delivery
Acronym: FORGE AHEAD
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Western Ontario, Canada (Other); First Nation Community Partners (Unknown); Health Canada (Other Government); First Nations and Inuit Health Branch (Unknown); Assembly of First Nations (Unknown); Canadian Diabetes Association (Other); Ontario Stroke Network (Other); Heart and Stroke Foundation of Canada (Other); Toronto Health Economics and Technology Assessment Collaborative (Unknown); Tri-Ethnic Research Center Colorado State University (Unknown); Hindsight Healthcare Strategies (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000031372
Record Dates: First submitted 2014-07-30; First posted 2014-09-09 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Quality Improvement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years

GROUPS / COHORTS (1):
- 11 First Nations Community and Clinical Teams: 11 Community & Clinical Teams in each First Nation community participated in the intervention.
  Interventions: Behavioral: Quality Improvement

INTERVENTIONS:
Behavioral: Quality Improvement — Community and Clinical Teams engaged in implementing Quality Improvement initiatives to improve diabetes prevention and management within their First Nations community and clinic.

SUMMARY:
Context: Indigenous peoples experience higher prevalence rates of diabetes and worse health outcomes compared to the general population because of a wide array of factors: social determinants of health, lifestyle, genetic susceptibility, and historic-political and psycho-social factors. Barriers to care that are unique to First Nations communities exacerbate the problem with fragmented healthcare, poor chronic disease management, healthcare staff turnover, and limited, or non-existent, surveillance.

Program: The TransFORmation of IndiGEnous PrimAry HEAlthcare Delivery (FORGE AHEAD) research program aims to develop and evaluate community-driven, culturally relevant, primary healthcare models that enhance chronic disease prevention and management in First Nations communities in Canada. Participants will consist of Indigenous community and clinic team members that will take part in multiple interrelated projects including community profiling, readiness consultations, diabetes registry and surveillance, and quality improvement workshops and action periods.

Design: This mixed-method pre-post observational study will capture: 1) diabetes clinical process and outcomes measures, 2) details about community-driven innovations, and 3) knowledge about the experience and cost of attempting to improve primary delivery in individual Indigenous communities.

Intervention/Instrument: Survey, literature review, 15 month intervention (readiness consultations, implementation and maintenance of a registry and surveillance system, community and clinic focused quality improvement workshops), interviews.

Measures: Primary- mean A1C of patients with diabetes (A1C ≥ 8.0% at baseline); Secondary-clinical process and outcome measures, change in stage of readiness, description of participation and innovation facilitators and barriers.

Policy Implications: The outcomes of this research program have the potential to significantly affect future policy decisions pertaining to chronic disease care in First Nations communities. Policy recommendations will be made to help support Indigenous communities in adopting successful innovations to help address issues related to diabetes and other chronic illnesses. The community-driven innovations developed in FORGE AHEAD and the subsequent policy decisions may enhance chronic disease prevention and management for Indigenous peoples across the country.

ELIGIBILITY:
Community members

Inclusion Criteria:

* 18 years of age or older
* on-reserve residents of participating Indigenous community partners

Exclusion Criteria:

* less than 18 years of age
* off-reserve residents of participating or non-participating Indigenous community partners

Clinic team members

Inclusion Criteria:

* Health centers of participating Indigenous community partners
* Current type 2 diabetes mellitus registry and surveillance system

Exclusion Criteria:

* Health centers of non-participating Indigenous community partners
* No registry or surveillance system

Diabetes Registry

Inclusion Criteria:

* adults (age≥ 18 years) with type 2 diabetes and most recent HbA1C≥ 8.0%

Exclusion Criteria:

* gestational diabetes, type 1 diabetes, or severe co-morbidity associated with life expectancy <6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Indigenous community and clinic team members
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
mean HbA1C of patients with diabetes (A1C ≥ 8.0% at baseline) | repeated measures: baseline (12 months prior to the start of the program)
mean HbA1C of patients with diabetes (A1C ≥ 8.0% at baseline) | repeated measures: 6 month after program start date
mean HbA1C of patients with diabetes (A1C ≥ 8.0% at baseline) | repeated measures: 12 month after program start date
mean HbA1C of patients with diabetes (A1C ≥ 8.0% at baseline) | repeated measure: 18 months after program start
mean HbA1C of patients with diabetes (A1C ≥ 8.0% at baseline) | repeated measure: 24 months after program start

CONTACTS AND LOCATIONS:
Overall Officials: Stewart B Harris, MD, MPH, Principal Investigator — Western University
Locations (1):
- Centre for Studies in Family Medicine, Western University, London, Ontario, Canada

REFERENCES:
- [Derived] Tompkins JW, Mequanint S, Barre DE, Fournie M, Green ME, Hanley AJ, Hayward MN, Zwarenstein M, Harris SB; FORGE AHEAD Program Team. National Survey of Indigenous primary healthcare capacity and delivery models in Canada: the TransFORmation of IndiGEnous PrimAry HEAlthcare delivery (FORGE AHEAD) community profile survey. BMC Health Serv Res. 2018 Nov 1;18(1):828. doi: 10.1186/s12913-018-3578-8. PMID 30382912
- [Derived] Hayward MN, Mequanint S, Paquette-Warren J, Bailie R, Chirila A, Dyck R, Green M, Hanley A, Tompkins J, Harris S; FORGE AHEAD Program Team. The FORGE AHEAD clinical readiness consultation tool: a validated tool to assess clinical readiness for chronic disease care mobilization in Canada's First Nations. BMC Health Serv Res. 2017 Mar 23;17(1):233. doi: 10.1186/s12913-017-2175-6. PMID 28335823
- [Derived] Naqshbandi Hayward M, Paquette-Warren J, Harris SB; FORGE AHEAD Program Team. Developing community-driven quality improvement initiatives to enhance chronic disease care in Indigenous communities in Canada: the FORGE AHEAD program protocol. Health Res Policy Syst. 2016 Jul 26;14(1):55. doi: 10.1186/s12961-016-0127-y. PMID 27456349
- See also: Related Info — https://www.uwo.ca/diabetesalliance/indigenous/forge_ahead/index.html?fbclid=IwAR0I2pLaNnglhcgRb_bWQwkMCIfY-SOLcgX_sDgoz2ydrnVnYdjDRUfLqZk